CLINICAL TRIAL: NCT03066089
Title: Open Labeled, Interventional, Two Armed, Single Centric Study to Assess the Efficacy of Fenfuro (Fenugreek Seed Extract) in Type-2 Diabetic Subjects: an add-on Study
Brief Title: Clinical Evaluation of Fenfuro (Fenugreek Seed Extract) in Type-2 Diabetic Subjects: an add-on Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-FEN/PREDIA/02/15
Record Dates: First submitted 2016-11-01; First posted 2017-02-28 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: FBS,HbA1C, PPBS
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — fenugreek seed meal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Fenfuro 500 mg capsule by mouth, BD (two times a day), till next follow-up
  Interventions: Drug: Fenfuro
- Group B (No Intervention): Investigational product is not being administered to this arm. This arm will regularly be observed on follow-up and laboratory investigations will be performed.

INTERVENTIONS:
Drug: Fenfuro
  Other Names: Fenugreek seed extract
  Arms: Group A

SUMMARY:
This study is an open label, two armed trial evaluating the safety and efficacy of Fenfuro capsule twice daily for 90 days in 100 patients with type 2 diabetes that will be conducted in single center in India. The primary outcome measures will be the determination of decrease in plasma glucose levels from baseline to last visit. The secondary outcome will be the determination of safety of Fenfuro capsule in type 2 diabetic subjects.

DETAILED DESCRIPTION:
Diabetes mellitus, involving rise in blood sugar levels, has shown to be a highly prevalent disease. Treatments and treatment regimens include combinations of oral anti-diabetic drugs (OADs), anti-hypertensive medications and anti-dyslipidemic agents, but these have been less than successful in managing their respective disease targets with clinical goals. Now-a-days, the treatment strategies for diabetes mellitus type 2 which are opted by general population include natural supplements. This choice is based upon the involvement of very less side effects along with high effectiveness of the natural supplements as compared to the synthetic medications. One of those natural supplements is fenugreek seeds extract i.e. Fenfuro which has been used as a nutraceutical in the present study for the management of type 2 diabetes mellitus.

Fenugreek has been extensively used as a source of anti-diabetic compounds from long time. Thus, Fenfuro, prepared from fenugreek seeds extract, is supposed to have anti-diabetic properties as well. Previous studies on fenugreek seeds extract have shown effective and safe anti-diabetic and anti-hyperlipidemic properties of it. It has shown to decrease blood glucose levels as well as lipid profile of the diabetic patients.

In this proposed study, Fenugreek seed extract will be used as an add-on to the existing therapy in patients with type-2 diabetes. The efficacy and safety of the extract will be evaluated using standard methodology.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to written as well as audio-visual informed consent.
* Patients of either sex.
* Aged 18-65 years.
* Fasting plasma glucose level <180 mg/dL.
* HbA1c level more than 7.5%.
* Not receiving any steroids.
* Patient on anti-diabetic therapy.

Exclusion Criteria:

* Uncooperative Subjects.
* Diabetes other than type-2 diabetes mellitus.
* Evidence of renal & liver disease.
* History of any hemoglobinopathy that may affect determination of HbA1c.
* Lactating and Pregnant or planning to conceive females.
* Physically/ mentally unwell as certified by physician-in-charge.
* Participation in any other clinical trial with in the last 30 days.
* Subjects with allergy to investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Blood Sugar | On completion of treatment (i.e.12 weeks) as compared to baseline
Change in Postprandial sugar | On completion of treatment (i.e.12 weeks) as compared to baseline

SECONDARY OUTCOMES:
Change in HbA1c levels | On completion of treatment (i.e.12 weeks) as compared to baseline
SGPT,SGOT,ALP,Creatinine,TLC,DLC & Hb | On completion of treatment (i.e.12 weeks) as compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Gian Sagar Medical College & Hospital, Rajpura, Punjab, India

IPD SHARING:
Plan to Share IPD: No